CLINICAL TRIAL: NCT00243048
Title: Phase II Randomized Study of Soy Isoflavones in Patients With Localized Prostate Cancer Treated With Radiation Therapy
Brief Title: Isoflavones and Radiation Therapy in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000446088; P30CA022453 (NIH); WSU-D-2325
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: soy protein isolate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Eating a diet high in soy foods may slow the progression of some types of cancer. Isoflavones are compounds found in soy food that may slow the growth of prostate cancer cells and prevent further development of prostate cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving isoflavones together with radiation therapy may be an effective treatment for prostate cancer.

PURPOSE: This randomized phase II trial is studying the side effects and how well giving isoflavones together with radiation therapy works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of soy protein isolate (isoflavones) and radiotherapy on the modulation of biomarkers in patients with localized prostate cancer.
* Determine the toxicity of this regimen in these patients.
* Determine the effect of this regimen on the quality of life of these patients.

OUTLINE: This is a randomized, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral soy protein isolate (isoflavones) twice daily for 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive an oral placebo twice daily for 6 months in the absence of disease progression or unacceptable toxicity.

In both arms, patients also undergo radiotherapy while receiving isoflavones or placebo.

Quality of life is assessed periodically.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate that is localized to the prostate gland
* Must be scheduled to receive curative radiotherapy for prostate cancer
* Not eligible for a higher priority study at the Karmanos Cancer Institute

PATIENT CHARACTERISTICS:

Performance status

* 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No organ function restrictions

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior hormonal therapy

Radiotherapy

* See Disease Characteristics

Other

* No other concurrent micronutrient supplements, herbs, or vitamins except 1 daily multivitamin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2002-05; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Oxidative DNA damage at 3 and 6 months

SECONDARY OUTCOMES:
Quality of life as measured by questionnaire at 3 and 6 months
Toxicity as measured by number and grade of adverse events weekly during radiation and at 3 and 6 months
Response as measured by prostate-specific antigen and clinical assessment at 3 and 6 months
Isoflavone serum level at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States